CLINICAL TRIAL: NCT05821101
Title: Clinical Outcomes of Clareon Vivity Intraocular Lens With Mini-Monovision Approach
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Debbie S. Kuo, MD (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Sponsor-Investigator, Debbie S. Kuo, MD, Ophthalmologist, Palo Alto Medical Foundation
Organization: Palo Alto Medical Foundation (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT# 76030963
Record Dates: First submitted 2023-04-07; First posted 2023-04-20 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-06

CONDITIONS: Aphakia, Postcataract
MeSH Terms: conditions — Aphakia, Postcataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Mini-Monovision Arm (Experimental): Bilateral implantation of Clareon Vivity and Clareon Vivity Toric IOLs targeted for mini-monovision.
  Interventions: Device: Clareon Vivity and Clareon Vivity Toric IOLs targeted for mini-monovision with dominant eye set at emmetropia and non-dominant eye at -0.50.

INTERVENTIONS:
Device: Clareon Vivity and Clareon Vivity Toric IOLs targeted for mini-monovision with dominant eye set at emmetropia and non-dominant eye at -0.50. — Bilateral implantation of IOLs such that dominant eye is corrected for distance vision while the non-dominant eye is corrected with a small amount of nearsightedness (-0.5 diopters).

SUMMARY:
Purpose is to study the clinical outcomes of Clareon Vivity and Clareon Vivity Toric intraocular lens (IOL) implants in patients who are planning to have cataract surgery in both eyes with a mini-monovision approach.

DETAILED DESCRIPTION:
A "mini-monovision" approach is one in which the dominant eye is corrected for distance vision while the non-dominant eye is corrected with a small amount of nearsightedness (-0.5 diopters). This approach can have the benefit of increasing ability to see over a broad range of vision without glasses. The Clareon Vivity and Vivity Toric lenses have been approved by the U.S. Food and Drug Administration (FDA) for visual correction of aphakia in adult patients following cataract surgery. It has lens technology that provides an extended depth of focus (more range of clear vision for distance, intermediate and near vision) compared to a standard monofocal (single focus) lens. None of the procedures in this study are experimental. However, the study is seeking additional information on clinical outcomes of the mini-monovision approach specifically using the Clareon Vivity and Vivity Toric lenses.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with bilateral age-related visually significant cataracts in otherwise healthy eyes, undergoing bilateral sequential implantation within 21 days using Clareon Vivity and Clareon Vivity Torics
* IOL powers between +10D to +30.0D, T3-T6
* Potential acuity measured post-operatively 20/25 or better in both eyes

Exclusion Criteria:

* History of ocular or refractive surgery
* Ocular or systemic comorbidities that may alter or reduce visual acuity, contrast sensitivity, binocularity, or impair reading performance such as severe dry eye/ocular surface disease, glaucoma, macular degeneration, retinopathy, neuro-ophthalmic diseases, strabismus/amblyopia etc.
* Patients with irregular astigmatism, corneal dystrophies, pupil abnormalities, zonular laxity
* Intraoperative or postoperative complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-04-06 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Binocular distance is target-corrected visual acuity (VA) at near 40cm. | 3 month post-surgery
  Increase in ability to see over a broad range of vision without glasses

CONTACTS AND LOCATIONS:
Locations (1):
- Palo Alto Medical Foundation, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No